CLINICAL TRIAL: NCT05942352
Title: Clinical Study of Ligustrazine in Treating Alcohol Addiction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Kangning Hospital (Other)
Responsible Party: Principal Investigator, Xiaojian Jia, Professor, Shenzhen Kangning Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-K003-02
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Abuse; Arteriosclerosis
Keywords: Alcohol; Addiction; Arteriosclerosis; Ligustrazine
MeSH Terms: conditions — Alcoholism; Arteriosclerosis; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Enrolled participants would accept intravenous administration of 250ml saline per day for 15 days, then 50 mg placebo tablet by mouth would be maintained for 1 year.
  Interventions: Drug: Placebo by intravenously administration; Drug: Placebo by mouth
- Ligustrazine short-term treatment (Experimental): Ligustrazine hydrochloride was administered intravenously by dissolving 40mg in 250ml saline per day for 15 days. Then, a 50 mg placebo tablet by mouth would be maintained for 1 year
  Interventions: Drug: Ligustrazine by intravenously administration; Drug: Placebo by mouth
- Ligustrazine maintenance treatment (Experimental): Ligustrazine hydrochloride was administered intravenously by dissolving 40mg in 250ml saline per day for 15 days，then, a 50 mg Ligustrazine tablet by mouth would be maintained for 1 year.
  Interventions: Drug: Ligustrazine by intravenously administration; Drug: Ligustrazine by mouth

INTERVENTIONS:
Drug: Ligustrazine by intravenously administration — Ligustrazine hydrochloride was administered intravenously by dissolving 40mg in 250ml saline per day for 15 days
  Other Names: Tetramethylpyrazine by intravenously administration
  Arms: Ligustrazine maintenance treatment; Ligustrazine short-term treatment
Drug: Ligustrazine by mouth — 50 mg Ligustrazine tablet by mouth would be maintained for 1 year
  Other Names: Tetramethylpyrazine by mouth
  Arms: Ligustrazine maintenance treatment
Drug: Placebo by intravenously administration — Intravenous administration of 250ml saline per day for 15 days
  Other Names: Saline by intravenously administration
  Arms: Placebo
Drug: Placebo by mouth — 50 mg placebo tablet by mouth would be maintained for 1 year
  Other Names: Starch tablet by mouth
  Arms: Ligustrazine short-term treatment; Placebo

SUMMARY:
Alcohol consumption is one of the most important risk factors for chronic non-communicable diseases in the population, and it is also the main cause of death from cancer, cardiovascular disease and lung disease, causing serious health, economic and social problems. The current alcohol-abstinence drugs have limited therapeutic effects and still present a high relapse rate. It is an urgent need to develop effective drugs for the treatment of alcohol addiction. The multimodal mechanism of action of ligustrazine in the central nervous system indicates that ligustrazine is expected to be developed as a potential therapeutic drug for alcohol addiction. Our study investigated the therapeutic effect of ligustrazine on subjects with alcohol addiction and the mechanism of multimodal brain imaging by administering ligustrazine, in order to develop new targeted drugs for alcohol treatment and provide more effective diagnosis and treatment methods for clinical treatment.

DETAILED DESCRIPTION:
Background: Alcohol use disorders (AUD) is a common chronic disease with great harm to society, causing a huge disease burden and social burden. In recent years, a lot of progress has been made in the field of drug abuse in the field of neurobiology, but it is difficult to apply it to AUD. The clinical treatment of alcohol addiction has always been under the predicament of lack of medicine and drugs, and the development of new therapeutic intervention methods is urgently needed. Although the neurobiological mechanism of ligustrazine's efficacy is still unclear, its multimodal mechanism of action in the central nervous system suggests that ligustrazine is expected to be developed as a potential therapeutic drug for alcohol addiction. Objective: This study intends to develop a therapeutic drug that can effectively relieve alcohol withdrawal syndrome, promote the disappearance of addictive behaviors, and effectively prevent re-drinking for the main active ingredient ligustrazine of the traditional Chinese medicine Ligusticum chuanxiong. The implementation of this project will help to expand the new functions (new indications) of traditional Chinese medicine and its main active ingredient ligustrazine, which may be developed into an effective drug for the treatment of alcohol addiction, and explore its neuroimaging mechanism. METHODS: Eligible alcohol addiction cases were recruited and assigned to 3 treatment groups according to randomized double-blind procedure (conventional treatment + placebo control group, conventional treatment + ligustrazine short-term treatment group, conventional treatment + ligustrazine maintenance treatment group ; about 100 cases in each group). After 15 days of group treatment, follow-up for 1 year, observe and compare the relapse rate of alcohol addiction, the duration of abstinence (days), the frequency and amount of drinking, the degree of craving, and other cognitive and psychological changes in each group, and record adverse reactions. Clinical efficacy and safety of ligustrazine on alcohol addiction. The changes of multimodal brain imaging in each group were analyzed, and the neural effects of ligustrazine treatment were explored. ②Recruit healthy controls ≥ 100 cases, match the sex and age with the cases, collect cognitive psychological indicators and brain imaging data at baseline and 1 year after baseline, and compare them in parallel with each treatment group to explore the treatment of alcohol addiction with Ligustrazine neural mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Alcohol addiction:

   ①Aged 18~65 years old;

   ② Meet the diagnostic criteria of DSM-IV alcohol dependence;

   ③No clear history of neurological diseases in the past, no family history of mental diseases;

   ④Voluntary participation in research, with good follow-up and observation, and good compliance;

   ⑤ No obvious psychotic symptoms.
2. Combined with the therapeutic indications of ligustrazine, selected cases must meet any of the following criteria on the premise of normal coagulation routine (no bleeding tendency): D-2 polymer ≥500 (thrombotic tendency) or atherosclerosis index ≥4 or one or more blood lipid indicators (TC, HDL, LDL) are abnormal.

Arteriosclerosis index (AI) = [total cholesterol (TC) - high-density lipoprotein (HDL)] ÷ high-density lipoprotein (HDL), the normal value of AI is <4, reflecting that the degree of arteriosclerosis is not serious or mild, The smaller the value, the lighter the degree of arteriosclerosis. If the arteriosclerosis index ≥ 4, it means that obvious arteriosclerosis has occurred, and the larger the value, the more serious the degree of arteriosclerosis.

Exclusion Criteria:

* ① Acute alcohol withdrawal phase, CIWA-Ar > 9 points;

  * Severe neurological or mental diseases caused by diseases other than chronic alcohol dependence: such as stroke, intracranial infection, brain tumor, schizophrenia, etc.;

    * Have experienced traumatic brain injury or other damage to brain tissue; ④ Taking any other psychotropic drugs, drug use or other substance dependence in the short term; ⑤ There are contraindications to the application of ligustrazine, or women are pregnant and other conditions that are not suitable for drug use; ⑥ There are conditions that are not suitable for head MRI examination, such as claustrophobia, metal objects in the body, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | Four week after treatment
  Percentage of participants who relapse by assuming that drinking alcohol on more than 3 days in a month in an unrestricted environment is re-drinking

SECONDARY OUTCOMES:
Time to maintain abstinence | Four week after treatment
  Measurement of exactly time(days) to maintain abstinence
Frequency of alcohol consumed | Four week after treatment
  Assessment of frequency to consume alcohol
Amount of alcohol consumed | Four week after treatment
  The amount of alcohol consumed would be measured.
Change from baseline in alcohol craving by using Visual Analog Scale of Alcohol Craving at week 4. | Four week after treatment
  Alcohol-specific Visual Analog Scale is a valid measurements of craving for a alcohol. Possible scores range from 0 (no craving) to 10 (want to drink imediately). Change= (week 4 score - baseline score)
Percent Mean Change in Blood Oxygen-level Dependent (BOLD) Scores | Four week after treatment
  BOLD fMRI signals evaluate different brain ROI

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojian Jia, Principal Investigator — Shenzhen Kangning Hospita
Locations (1):
- Shenzhen Kangning Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
not decided